CLINICAL TRIAL: NCT01093092
Title: A Phase I Clinical Trial of Oral Calcitriol With Fixed Dose of Cisplatin and Gemcitabine in Patients With Advanced Solid Tumors
Brief Title: Calcitriol, Cisplatin, and Gemcitabine Hydrochloride in Treating Patients With Advanced Solid Tumors That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study transferring to INOVA Health
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 163509; NCI-2010-00263 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 163509 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — Calcitriol; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (calcitriol, cisplatin, gemcitabine hydrochloride) (Experimental): Patients receive calcitriol PO on days 1, 2, 8, 9, 15 and 16; cisplatin IV over 2 hours on day 2; and gemcitabine hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Calcitriol; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Dietary Supplement: Calcitriol — Given PO
  Other Names: 1,25(OH)2-D3; 1,25-Dihydroxycholecalciferol; Calcijex; Rocaltrol
Drug: Cisplatin — Given IV
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of calcitriol when given with cisplatin and gemcitabine hydrochloride in treating patients with advanced solid tumors that cannot be removed by surgery. Drugs used in chemotherapy, such as cisplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Calcitriol may stop the growth of tumor cells by blocking blood flow to the tumor. Calcitriol may also help cisplatin and gemcitabine hydrochloride kill more tumor cells by making them more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of oral calcitriol when combined with a standard dose of gemcitabine (gemcitabine hydrochloride) and cisplatin in a 28-day cycle.

SECONDARY OBJECTIVES:

I. Describe the toxicity of this combination using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

II. Study the pharmacokinetics of calcitriol at the maximum tolerated dose (MTD) in an expanded cohort of 6 patients.

III. Describe the clinical activity associated with this regimen in this advanced solid tumor population.

OUTLINE:

Patients receive calcitriol orally (PO) on days 1, 2, 8, 9, 15 and 16; cisplatin intravenously (IV) over 2 hours on day 2; and gemcitabine hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of advanced unresectable non-hematological malignancy that has no known standard of care or for which the use of gemcitabine plus cisplatin constitutes a reasonable option
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* White blood cell (WBC) >= 3.0 x 10^9/L
* Neutrophils >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hgb) >= 10 g/dL
* Bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x institutional ULN unless metastatic to liver in which case AST and ALT should be < 5 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Corrected calcium =< institutional ULN (corrected calcium = (4- Albumin) x 0.8 + calcium)
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* No treatment with investigational agents within 4 weeks prior to study drug administration, except patients receiving targeted therapies such as kinase inhibitors with half-lives < 48 hours may be treated if > 14 days have elapsed after the last dose and related toxicities have recovered to =< grade 1
* No chemotherapy within 4 weeks prior to study treatment administration; nitrosoureas and mitomycin C are not allowed within 6 weeks prior to initiation of study treatment
* Palliative radiation, including whole brain radiation therapy (WBRT), is allowed prior to enrollment as long as it is completed > 2 weeks from initiation of study treatment, and provided patient has recovered from treatment toxicities to =< grade 1
* Patients should be able to take oral medications

Exclusion Criteria:

* Known hypersensitivity to any of the study drugs involved
* Brain metastases are excluded unless treated and shown to be controlled more than 1 month from after craniotomy or more than 2 weeks after gamma knife radiosurgery and not associated with central nervous system (CNS) symptoms
* History of clinically significant hypercalcemia
* Evidence of nephrectomy
* History of (within 24 months prior to enrollment) of kidney, ureter, or bladder stones with clinically significant sequelae (e.g. (painless gross hematuria; pain with or without infection; hydronephrosis, etc); patients with otherwise stable non-occluding kidney stones regardless of stone type incidentally found in computed tomography (CT) scans are eligible; patients with prior history of uric acid stones are eligible regardless of time of onset
* Unwillingness to stop calcium supplementation (during the first cycle of treatment) or vitamin D supplementation throughout the study
* Thiazide (e.g HCTZ, Hydrochoirthiazide) or digoxin therapy (e.g Lanoxicaps, Lanoxin)
* Pregnant or nursing female patients.
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 4 weeks prior to enrollment, except patients receiving targeted therapies such as kinase inhibitors with half-lives < 48 hours may be treated if > 14 days have elapsed after the last dose and related toxicities have recovered to =< grade 1
* Nut allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
MTD of oral calcitriol when combined with a standard dose of gemcitabine hydrochloride and cisplatin, determined according to incidence of dose-limiting toxicity, graded using the National Cancer Institute (NCI) CTCAE version 4.0 | 28 days
  A standard 3+3 with de-escalation will be used to estimate the MTD.

SECONDARY OUTCOMES:
Toxicity of this combination, graded according to NCI CTCAE version 4.0 | Up to 30 days after last dose of study drug
  Tabulated overall or by dose level (as appropriate).
Pharmacokinetic (PK) analyses of calcitriol at the MTD in an expanded cohort of 6 patients, including peak levels, area under the concentration-time curve from time 0-72 hours, terminal half-life, volume of distribution, and total body clearance | Days 1-3 of course 1
  PK data will be presented as plots of serum calcitriol concentration over time for each patient. An assessment of whether systemic calcitriol exposure associated with antitumor activity in preclinical models is achieved in these patients will be made.
Objective tumor response, described using Response Evaluation Criteria in Solid Tumors 1.1 | Up to 5 years
  Responses tabulated as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Dy, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia